CLINICAL TRIAL: NCT06502405
Title: Research on the Application of Electrical Impedance Tomography in Bronchial Challenge Testing
Status: Not yet recruiting | Type: Observational
Sponsor: wang kaifei (Other)
Responsible Party: Sponsor-Investigator, wang kaifei, Deputy chief physician, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: EIT and PFTs
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to examine whether electrical impedance tomography (EIT) was capable of identifying the deteriorated lung function on a regional level during bronchial challenge testing and whether EIT may provide additional information during bronchial challenge testing and identify spatial and temporal heterogeneity of regional lung function.

DETAILED DESCRIPTION:
The content of this study includes:

1. Can EIT identify the uneven ventilation caused by airway contraction in patients during bronchial provocation tests.
2. Can EIT monitor airway contraction in patients before Spirometer examination after inhaling activators.
3. Can EIT observe uneven ventilation caused by airway contraction through tidal breathing after the patient inhales activator.

ELIGIBILITY:
Inclusion Criteria：

1. Patients suspected of asthma who require bronchial challenge testing.
2. The Bronchodilator responsiveness testing is negative.
3. patients with a pre-bronchodilator FEV1 >60% predicted.
4. No contraindications for bronchial provocation test examination.
5. Fully understand the purpose and significance of this study, and voluntarily participate in the research.

Exclusion Criteria:

1. patients with a pre-bronchodilator FEV1≤60% predicted.

1. Contraindications for bronchial challenge testing.
2. Pregnant or lactating women.
3. After pacemaker surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients need to exclude or confirm a suspected diagnosis of asthma through bronchial challenge testing.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
global inhomogeneity index （GI） | 1day
  Measured by EIT, used to describe the overall degree of spatial heterogeneity of ventilation.
forced expiratory volume in 1s (FEV1) | 1day
  The forced expiratory volume in 1s measured during pulmonary function tests.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Xie, Dr, Study Director — Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and research data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 1 year after the publication of research results.
Access Criteria: Can be obtained from the main researcher.